CLINICAL TRIAL: NCT03625557
Title: Guardant360® Test-Related Clinical Outcomes in Patients Who Share Medical Records (GRECO)
Brief Title: Guardant360® Test-Related Clinical Outcomes in Patients Who Share Medical Records
Status: Completed | Type: Observational
Sponsor: Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 01-MX-002
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Non-Hematologic Malignancy
Keywords: Guardant Health; GRECO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To document the clinical outcomes of cancer patients who received the Guardant360® test and agree to share their records with Guardant Health.

DETAILED DESCRIPTION:
This is an observational study of clinical outcomes to be conducted in the United States. Patients with a diagnosis of Stage 3-4 advanced cancer who possess specific pathway mutations identified by the Guardant360® test will be eligible to enroll in the study. Patients will be recruited by telephone or email and/or through the Guardant Health Patient Portal to determine interest in the study. Should patients be interested in contributing to this registry study, they will be prompted to consent via a commercial service for patients to request, manage, and view their medical records. Enrolled participants will be requested to release copies of their medical records for review by the principal investigator. Study adminsitrators will abstract participant demographics, cancer-related therapies, and clinical outcomes for analysis.

ELIGIBILITY:
General Inclusion Criteria:

* Adults (≥ 18 years old) with a diagnosis of Stage 3 or Stage 4 cancer (non-hematologic malignancy). Patients with advanced cancers not typically staged 1-4 (such as extensive stage small lung cancer) may be enrolled.
* Results from Guardant360® test
* Patient has previously provided contact information (either email or phone) to Guardant Health.
* Able and wiling to complete the informed consent process.
* Willingness to consent to the release of medical records.
* Willingness to provide Medical Records Release

General Exclusion Criteria:

* Unwilling or unable to provide written informed consent.
* Unable to understand English.
* Diagnosis of NSCLC
* Guardant 360® test results released to the patient's physician no less than 14 days and no greater than 60 days prior to initial patient contact.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with advanced cancer involving genetic pathway alterations identified through Guardant 360®.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 years
  Portion of patients with tumors that are found to have complete or partial response

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Lang, MBBS, MRCP, FRCPath, Principal Investigator — Guardant Health, Inc.
Locations (1):
- Guardant Health, Redwood City, California, United States